CLINICAL TRIAL: NCT00967980
Title: Femoral Versus Psoas Continuous Peripheral Nerve Blocks Following Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Dr. Brian Ilfeld, University of California, San Diego, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Femoral vs. Psoas PNB Cath Hip
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Hip Arthroplasty; Hip Pain
Keywords: pain; Hip Resurfacing; catheter; nerve block; UCSD; hip surgery; psoas; femoral; ambulation; hip flexion; infusion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Femoral Nerve Block (Active Comparator): Patients will be randomized with a computer program to receive a femoral catheter. The catheter will be placed using standard technique. The time of catheter placement will be recorded as well as the pain/discomfort of catheter placement as reported by the patient on a 0-10 scale where 0=no pain/discomfort and 10=worst imaginable pain/discomfort.
  Interventions: Procedure: Femoral Nerve Block vs. Psoas Compartment Nerve Block
- 2. Psoas Compartment Catheter (Active Comparator): Patients will be randomized with a computer program to receive a psoas compartment catheter. The catheter will be placed using standard technique. The time of catheter placement will be recorded as well as the pain/discomfort of catheter placement as reported by the patient on a 0-10 scale where 0=no pain/discomfort and 10=worst imaginable pain/discomfort.
  Interventions: Procedure: Femoral Nerve Block vs. Psoas Compartment Nerve Block

INTERVENTIONS:
Procedure: Femoral Nerve Block vs. Psoas Compartment Nerve Block — Patients, undergoing hip arthroplasty or hip resurfacing will be randomized to one of two groups: femoral nerve block or psoas compartment nerve block. Patients randomized to femoral nerve block will receive this block prior to surgery. Patients randomized to psoas compartment nerve block will receive this block prior to surgery. Both patients will receive Mepivicaine via catheter prior to surgery and following surgery, Ropivicaine via pain pump.

SUMMARY:
The purpose of this research study is to determine if the insertion site of a perineural catheter, or tiny tube placed next to the nerves that go to the hip which you will have surgery, affects the amount of pain relief that is experienced after surgery.

DETAILED DESCRIPTION:
To determine the association between perineural catheter location and postoperative analgesia, analgesic requirements, ambulatory distance, and flexion following hip arthroplasty.

Primary Hypothesis: Differing the catheter insertion site (femoral vs. psoas compartment) for a perineural local anesthetic infusion is not associated with lower pain scores during the 24-hour period beginning the morning following hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* primary, unilateral hip arthroplasty or hip resurfacing
* age greater than or equal to 18 years
* postoperative analgesic plan includes perineural local anesthetic infusion

Exclusion Criteria:

* morbid obesity (BMI greater than 40)
* chronic, high-dose opioid use
* history of opioid abuse
* pregnancy
* incarceration
* amu meirp-muscular deficit of the ipsilateral femoral nerve and/or quadriceps muscle
* inability to communicate with hospital staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Patient's mean pain score (NRS) during perineural infusion as measured by the nursing staff at UCSD and entered in the computer system. | 24 hours beginning 7:30am day following surgery

SECONDARY OUTCOMES:
Analgesic used, as reported by nursing staff in the UCSD computer system. | 3 days following surgery
Patient's ambulation distance as recorded by therapist (occupational or physical) in the UCSD computer system. | 3 days following surgery
Hip flexion, in degrees measured with a standard goneometer, as recorded by therapist (occupational or physical) in the UCSD computer system. | 3 days following surgery
Infusion duration of pain pump, measured on the pump itself in hours and minutes. | 3 days following surgery
Duration of hospital stay, in hours, as reported in the UCSD computer system. | 3 days following surgery
Surgical/anesthetic adverse events as reported by hospital staff | day of surgery and 3 days following
Experiences of patient during the infusion and following, as reported to study staff in a phone conversation, one week following surgery. | 1 week following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

REFERENCES:
- [Derived] Ilfeld BM, Mariano ER, Madison SJ, Loland VJ, Sandhu NS, Suresh PJ, Bishop ML, Kim TE, Donohue MC, Kulidjian AA, Ball ST. Continuous femoral versus posterior lumbar plexus nerve blocks for analgesia after hip arthroplasty: a randomized, controlled study. Anesth Analg. 2011 Oct;113(4):897-903. doi: 10.1213/ANE.0b013e318212495b. Epub 2011 Apr 5. PMID 21467563